CLINICAL TRIAL: NCT00697827
Title: A Multi-Center Randomized Controlled Trial of the In-Space Compared to X STOP® for Treatment of Moderate Degenerative Lumbar Spinal Stenosis
Brief Title: A Study of the In-Space Device for Treatment of Moderate Spinal Stenosis
Acronym: In-Space
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to low enrollment.
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSP01
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Results first posted 2012-06-05 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): In-Space
  Interventions: Device: Interspinous Spacer device
- 2 (Active Comparator): X STOP
  Interventions: Device: Interspinous Process Distraction Device

INTERVENTIONS:
Device: Interspinous Spacer device — Device: In-Space
  Arms: 1
Device: Interspinous Process Distraction Device — Device: X STOP
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the In-Space compared to the X STOP Interspinous Process Distraction (IPD) device ("X STOP") for the treatment of patients experiencing intermittent neurogenic claudication secondary to moderate degenerative lumbar stenosis at one or two lumbar levels.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years in age
* Leg/buttock/groin pain, with or without back pain, that can be completely relieved by flexion such as when sitting in a chair.
* Zurich Claudication Questionnaire Score ≥ 2.0,
* Neurogenic intermittent claudication secondary to moderate lumbar spinal stenosis
* Has completed at least 6 months conservative therapy

Exclusion Criteria:

* Axial back pain only without leg/buttock/groin pain
* Has had any prior lumbar spine surgery at any level
* Significant scoliosis, defined as Cobb angle > 10°
* Spondylolisthesis > Grade 1 or isthmic spondylolisthesis at affected level
* Osteoporosis
* Morbid obesity, defined as BMI > 40 kg/m2

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - The Spine Institute, Santa Monica, California
  - Yale Orthopedics, New Haven, Connecticut
  - Institute for Low Back and Neck Care, Minneapolis, Minnesota
  - Cornell University Hospital, New York, New York
  - OrthoCarolina Spine Center, Charlotte, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Neurosurgical Associates at Centennial Medical Center, Nashville, Tennessee
  - Texas Back Institute, Plano, Texas
  - Neurosurgical Specialists, Inc., Norfolk, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- In-Space: The treatment group consists of patients who receive the In-Space device. The In-Space is indicated for patients experiencing intermittent neurogenic claudication secondary to degenerative lumbar stenosis. Moderate degenerative lumbar stenosis is further defined by moderately impaired physical function in patients who experience relief in flexion from their symptoms of leg/buttock/groin pain, with or without back pain, and have undergone a regimen of at least 6 months of conservative treatment, and who otherwise would not be treated by a surgical decompression. The In-Space is intended to be implanted between the spinous processes of 1 or 2 contiguous lumbar motion segments between L1 and L5.
- X-Stop: The control group consists of patients who receive X STOP which is an appropriate control as the X STOP is FDA-approved. The X-Stop Interspinous Process device is indicated for treatment of patients aged 50 or older suffering from neurogenic intermittent claudication secondary to a confirmed diagnosis of lumbar spinal stenosis. The X-Stop may be implanted at one or two lumbar levels in patients in whom operative treatment is indicated at no more than two levels.
Period: Overall Study
Arm/Group | In-Space | X-Stop
Started | 28 | 16
Completed | 26 | 15
Not Completed | 2 | 1
Not completed — enrolled but not treated | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Space | X-Stop | Total
Number analyzed (Participants) | 28 | 16 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 7 | 23
  >=65 years | 12 | 9 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 63.1 (7.88) | 64.8 (6.69) | 64.0 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 25
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 28 | 16 | 44

OUTCOME MEASURES:

1. Primary Outcome: Zurich Claudication Questionnaire(ZCQ)
Description: The questionnaire quantifies severity of symptoms, physical function characteristics, and patient's satisfaction. The scale relates to symptoms over the past month. The result is expressed as a percentage of the maximum possible score. The score increases with worsening disability. An individual patient treatment will be considered a success if they meet at least two of three components defined as an improvement of ≥ 0.5 as compared to preoperative score for the symptom severity and physical function and an of < 2.5 points for patient satisfaction at 24 months.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | In-Space | X-Stop
Number analyzed (Participants) | 26 | 15
participants | 17 | 7

2. Secondary Outcome: Oswestry Disability Index (ODI)
Description: The Oswestry Disability Index (ODI) is one of the principal condition-specific outcome measures used in the management of spinal disorders. There are 10 questions. The questions are designed in a way to show how the back or leg pain is affecting the patient's ability to manage in everyday life. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score. For this study,any improvement at 24 months compared to pre-operative baseline was determined as a success.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | In-Space | X-Stop
Number analyzed (Participants) | 26 | 15
participants | 18 [0 to 60] | 6

ADVERSE EVENTS:
Arm/Group | In-Space | X-Stop
Serious Adverse Events (participants affected / at risk) | 19/28 | 9/16
Other Adverse Events (participants affected / at risk) | 21/28 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Space (N=28) | X-Stop (N=16)
Cardiovascular (Cardiac disorders) | 0 (0) | 1 (1)
Fracture Spine - not Spinous Process (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Back and Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Index Level Surgery (Surgical and medical procedures) | 5 (6) | 4 (4)
Surgery - not Index Level (Surgical and medical procedures) | 10 (18) | 4 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Space (N=28) | X-Stop (N=16)
Spinous Process Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Non-spine Fractures (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 4 (4) | 0 (0)
Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (2) | 0 (0)
Non-wound related Infection (Infections and infestations) | 1 (1) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal spasms back (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neurological (Nervous system disorders) | 2 (2) | 1 (1)
Numbness non-index level related (Nervous system disorders) | 1 (1) | 0 (0)
Other (General disorders) | 4 (8) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 3 (3)
Pain - back and other (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Pain - incision site (General disorders) | 1 (1) | 0 (0)
Pain - lower extremities (Musculoskeletal and connective tissue disorders) | 7 (12) | 5 (9)
Pain - neck (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain - neck and other (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3)
Pain - other (General disorders) | 3 (3) | 0 (0)
Pain - shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Psychological (Psychiatric disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Wound issues other (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Study terminated early secondary to low enrollment leading to small number of subjects available for analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All unpublished information given to the investigator by Synthes Spine shall not be published or disclosed to a third party without the prior written consent of Synthes Spine. All information concerning In-Space, Synthes Spine operations, patent application drawings, manufacturing processes, basic scientific data and design information, supplied by the sponsor to the investigator and not previously published, is considered confidential and remains the sole property of Synthes Spine.